CLINICAL TRIAL: NCT07020559
Title: Comparing Allogeneic Versus Autologous Platelet-Rich Plasma for Diabetic Wound Healing in Patients With Renal Dysfunction：a Randomized Controlled Trial
Brief Title: Allogeneic vs Autologous PRP for Diabetic Wounds in Renal Dysfunction: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Head of Wound Healing Center, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Long2025-DW-alPRP
Record Dates: First submitted 2025-06-06; First posted 2025-06-13 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Wounds; Platelet Rich Plasma; Allogeneic Blood Transfusions; Renal Dysfunction
Keywords: Diabetic wounds; Platelet Rich Plasma; allogeneic blood; renal dysfunction
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autologous platelet plasma group (Active Comparator): diabetic-related wounds after wound bed preparation are treated by the autologous platelet plasma
  Interventions: Drug: autologous platelet plasma
- allogeneic platelet plasma group (Experimental): diabetic-related wounds after wound bed preparation are treated by the allogeneic platelet plasma
  Interventions: Drug: allogeneic platelet plasma

INTERVENTIONS:
Drug: allogeneic platelet plasma — Al-PRP derived from healthy blood donors
  Arms: allogeneic platelet plasma group
Drug: autologous platelet plasma — Autologous platelet-rich plasma from the patient themselves
  Arms: autologous platelet plasma group

SUMMARY:
Diabetic wounds are difficult to heal. Autologous platelets in diabetic patients with renal insufficiency have poor function. Allogeneic platelet plasma has a promising application prospect. Comparing the efficacy and safety differences between allogeneic platelet plasma and autologous platelet plasma is of significant importance and value for the clinical application.

DETAILED DESCRIPTION:
This study is a single-center, randomized, parallel control, superior trial. Fifty-six renal dysfunction patients with diabetic-related wound after wound bed preparation will be randomly assigned to the autologous platelet plasma group and allogeneic platelet plasma group in a 1:1 ratio. The primary outcome is the wound healing rate at 4 weeks (Stitches removal). The secondary outcomes include the wound healing rates at 3 weeks, the reduction rate of wound area at 2-, 3- and 4- weeks, healing time, post-operative wound infection, 7-day, 2-, 3-, 4-week pain relief progression assessed by Visual Analog Scale, incidence of mortality, reoperation, and adverse events during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is aged 18-80 years old;
2. Diagnosed as type 1 or type 2 diabetes according to the World Health Organization standard, blood sugar has been controlled before enrollment, and the level of Glycated hemoglobin HbA1c is less than 10%;
3. Abnormal renal function defined as:

   * Serum creatinine >106 μmol/L (men) or >97 μmol/L (women)
   * AND eGFR <90 mL/min/1.73m² (CKD-EPI) ；
4. The patient has diabetes wounds with poor healing or prolonged healing need standard wound treatment;
5. After preparing the wound bed, the condition for using platelet plasma to close the wound is met*;
6. Voluntarily sign an informed consent form;

Exclusion Criteria:

1. Blood glucose is out of control or not yet effectively controlled，;
2. Severe diseases such as acute myocardial infarction, heart failure, hepatitis, shock, and respiratory failure have not been corrected yet;
3. Active bleeding inside the wound, and routine basic treatment plans cannot be implemented；
4. Uncontrolled systemic or disseminated infections;
5. Patients with advanced malignant tumors;
6. Pregnant or lactating women；
7. The patient is unable to cooperate or has mental disorders;
8. According to the judgment of the researchers, the patient has a clear and irremovable cause that affects wound healing, which is not suitable for this study or cannot comply with the requirements of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
the wound healing rate at 4 weeks | by the end of 4 weeks
  calculated as the percentage of healed wounds by the end of 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided